CLINICAL TRIAL: NCT06360692
Title: Impact of Nipple Micropigmentation in Mastectomized Women. Quasi-experimental Study
Brief Title: Impact of Nipple Micropigmentation in Mastectomized Women
Status: Not yet recruiting | Type: Observational
Sponsor: Cardenal Herrera University (Other)
Responsible Party: Principal Investigator, Marta Lluesma Vidal, assistant research scientist, Cardenal Herrera University
Other Study IDs: Marta Lluesma Vidal Carden
Record Dates: First submitted 2024-03-08; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Body Image; Female Sexual Function; Self Esteem; Intimacy With Your Partner
Keywords: breast cancer; nipple tattoing,; micropigmentation
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This will be a multicenter prospective descriptive case series study following a cohort.

The micropigmentation/tattoo procedure will be carried out following the protocol established in each center (see annex x). The present investigation only involves measuring the impact that this technique has on the patients by collecting data in digital format before and after the CAP micropigmentation/tattoo that motivated their visit to the clinical service.

CAP micropigmentation/tattooing is usually performed between 6 and 12 months after the breast reconstructive surgery has been completed, sufficient time for healing to complete and the breast to stabilize, although it can be performed from 2 months after the intervention. Nurses are responsible for performing micropigmentation/tattooing of the areola and nipple in mastectomized women.

DETAILED DESCRIPTION:
The micropigmentation/tattoo procedure will be carried out following the protocol established in each center. This research only involves measuring the impact that this technique has on patients by collecting data in digital format before and after micropigmentation/tattoo.

On the first visit, the patient is informed of the micropigmentation/tattoo technique, its benefits and possible side effects.

If the patient meets the eligibility criteria, the study will be explained to her and she will be asked to sign consent to participate in the study.

In addition, a first assessment of the skin is performed and the design that will be made is explained to the patient. During this first visit, the allergy test is performed, which consists of a minimal injection of pigment in the area where the tattoo will be done. All information is given to the patient in writing and on this occasion the patient signs the informed consent document to consent to this technique being performed. In this visit, data collection corresponding to T0 is carried out. To do this, you will be provided with a QR code that will allow you to access the battery of questionnaires that make up the data collection. In addition, the nurse will complete some of the clinical variables when the patient accesses said link.

Starting the week following the allergy test, the patient can be scheduled for the second visit, and if there is no allergy to the pigment, the micropigmentation/tattoo will be performed after designing the shape, size and color following the hospital's protocol.

The patient will be scheduled again for the micropigmentation/reconstructive tattoo consultation after a month and a half for review and assessment of the need for micropigmentation touch-up.

For the collection of T1 and T2 data, digital notifications will be programmed that will be sent automatically after 3 and 12 months with the link to access the battery of questionnaires. Telephone follow-up will be carried out to avoid losses.

The participants will be evaluated in three times:

T0: baseline measurement at the time of recruitment in the visit with the nurse performing the intervention coinciding with the scheduled appointment for the allergy test.

T1: measurement 3 months after micropigmentation/tattoo. Changes in body image are integrated after 4 weeks17 after any treatment or intervention.

T2: measurement one year after micropigmentation/tattoo.

ELIGIBILITY:
Inclusion Criteria:

* Having undergone a mastectomy and subsequent breast reconstruction as a result of breast cancer.
* Be able to read and understand the Spanish language.
* Have access to the internet

Exclusion Criteria:

* women who have previously had a nipple tattoo;
* women who refuse to participate in the study;
* pregnant or breastfeeding women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women undergoing micropigmentation of the areola-nipple complex in mastectomized patients who have undergone breast reconstruction treated in the following services: Plastic Surgery of the General University Hospital of Valencia (Spain), the Breast Micropigmentation Unit of the Puerta del Hierro Hospital in Madrid (Spain) and the Breast Surgery consultation at the San Juan Hospital in Alicante (Spain).
  Enviar comentarios
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Body imagen | base, 3 months, 12 months
  Hopwood Body Image Scale (BIS). Validated in Spanish by Gómez-Campelo & Bragado-Álvarez. This questionnaire presents Cronbach's alpha of 0.84 in the internal consistency analysis for Latina women with breast cancer and 0.93 in the general Spanish population. The questionnaire consists of 10 items that evaluate several dimensions of body image in cancer patients: affective, behavioral and cognitive. Items are scored on a four-point scale (0=not at all, 1=a little, 2=quite a bit, 3=a lot). The total score is the sum of the 10 items and ranges between 0 and 30. Higher scores correspond to a negative body image. The BIS is a brief, easy self-report instrument that is applicable to patients with any type of cancer, stage of disease, or treatment. Its use has increased in recent years, becoming a reference measure in international research.

SECONDARY OUTCOMES:
Self-esteem | base, 3 months, 12 months
  Rosenberg Self-esteem scale. Validated in Spanish by Morejón et al.. This questionnaire has a Cronbach's alpha coefficient of 0.89 and a two-week test-retest correlation coefficient of 0.91 for the Spanish population. This questionnaire consists of a scale of 10 items whose contents focus on feelings of respect and acceptance of oneself, of which 5 are written positively and 5 negatively with a 4-point Likert-type response format. according to the degree of agreement: 1 (strongly disagree), 2 (disagree), 3 (agree), 4 (strongly agree). To correct it, the scores of the negatively stated items must be reversed (3,5,8,9,10) and all the items must subsequently be added. The total score, therefore, ranges between 10 and 40.
Sexual Function | base, 3 months, 12 months
  Female sexual function index (FSFI), developed by Rosen et al. The questionnaire is validated in Spanish, showing good reliability with Cronbach's alpha (α) of 0.7. It is a questionnaire of 19 questions, grouped into six domains: desire, arousal, lubrication, orgasm, satisfaction and pain. Each question has 5 or 6 response options, assigning them a score ranging from 0 to 5. The total value of each domain is multiplied by a coefficient and the final result is the arithmetic sum of the domains. The higher the score, the better sexuality. It is a self-administered, simple and reliable questionnaire to evaluate female sexual function in a wide age range.
Intimacy with the partner | base, 3 months, 12 months
  Sexual Interaction Inventory (SII). Validated into Spanish by Aluja. In calculating reliability, Cronbach's alpha values (α) were obtained for the total scale between 0.79 and 0.93. The test-retest reliability at two weeks was between 0.5 and 0.9. It is a self-administered questionnaire whose objective is to evaluate the satisfaction and adjustment of a heterosexual couple. Only the first three items of the questionnaire will be used to assess the real and ideal frequency of each behavior, the degree of pleasure it provides to oneself and to the partner, as well as the degree of pleasure that you would like it to provide them.

CONTACTS AND LOCATIONS:
Overall Officials: Marta Lluesma-Vidal, Ph.D, Principal Investigator — CEU-Cardenal Herrera University, CEU universities

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hopwood P, Fletcher I, Lee A, Al Ghazal S. A body image scale for use with cancer patients. Eur J Cancer. 2001 Jan;37(2):189-97. doi: 10.1016/s0959-8049(00)00353-1. PMID 11166145
- [Background] Gomez-Campelo P, Bragado-Alvarez C, Hernandez-Lloreda MJ, Sanchez-Bernardos ML. The Spanish version of the Body Image Scale (S-BIS): psychometric properties in a sample of breast and gynaecological cancer patients. Support Care Cancer. 2015 Feb;23(2):473-81. doi: 10.1007/s00520-014-2383-0. Epub 2014 Aug 19. PMID 25135839
- [Background] Banos RM, Guillen V. Psychometric characteristics in normal and social phobic samples for a Spanish version of the Rosenberg Self-Esteem Scale. Psychol Rep. 2000 Aug;87(1):269-74. doi: 10.2466/pr0.2000.87.1.269. PMID 11026424
- [Background] Valenzuela-Peters R, Contreras-Garcia Y, Manriquez-Vidal C. Influence of the type of work shift in Female Sexual Function Index of healthcare sector female workers. Eur J Obstet Gynecol Reprod Biol. 2017 Mar;210:39-44. doi: 10.1016/j.ejogrb.2016.12.001. Epub 2016 Dec 6. PMID 27940265
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Background] Sanchez-Sanchez B, Navarro-Brazalez B, Arranz-Martin B, Sanchez-Mendez O, de la Rosa-Diaz I, Torres-Lacomba M. The Female Sexual Function Index: Transculturally Adaptation and Psychometric Validation in Spanish Women. Int J Environ Res Public Health. 2020 Feb 5;17(3):994. doi: 10.3390/ijerph17030994. PMID 32033334
- [Background] Morokoff PJ, LoPiccolo J. A comparative evaluation of minimal therapist contact and 15-session treatment for female orgasmic dysfunction. J Consult Clin Psychol. 1986 Jun;54(3):294-300. doi: 10.1037//0022-006x.54.3.294. No abstract available. PMID 3722555